CLINICAL TRIAL: NCT03746535
Title: Mechanisms and Interventions Addressing Accelerated Cardiovascular Disease Risk in Women With Endometriosis
Brief Title: Cardiovascular Disease Risk in Women With Endometriosis
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2000022193; 1R01HL161000-01 (NIH)
Record Dates: First submitted 2018-10-17; First posted 2018-11-19 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis | interventions — elagolix

STUDY DESIGN:
Intervention Model Description: 2 cohort clinical trial
Masking Description: no masking, all subjects have endometriosis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- patients without endometriosis (Active Comparator): Control subjects will be healthy women, with regular menses every 26-34 days. Subjects will be excluded if they have any symptoms of endometriosis, including severe dysmenorrhea or progressive cyclic pelvic pain or prior surgery showing evidence of endometriosis
  Interventions: Drug: Elagolix
- patients with endometriosis (Experimental): Endometriosis will be diagnosed by history of the disease seen at the time of prior surgery or will be diagnosed by classic clinical symptoms of the disease (cyclic progressive pelvic pain) using prior surgical report reviewed by Dr. Taylor.
  Interventions: Drug: Elagolix

INTERVENTIONS:
Drug: Elagolix — Elagolix, 400 mg/day oral, 2X200 mg tablets/day for 4 days.

SUMMARY:
To test the hypothesis that estrogen suppression impairs endothelial dysfunction in endometriosis.

DETAILED DESCRIPTION:
Our scientific premise is that in women with endometriosis, elevated cardiovascular disease risk is the result of endothelial dysfunction and chronic systemic inflammation through lectin-like oxidized low-density lipoprotein receptor-1 (LOX-1) receptor activation. This cardiovascular disease risk is exacerbated by standard estrogen suppression treatments.

ELIGIBILITY:
Inclusion Criteria:

* Young women between the ages of 18 and 45 years (Controls);
* Young women between the ages of 18 and 45 years with endometriosis.

Exclusion Criteria:

* Subjects who smoke
* Subjects who have diabetes,
* Subjects with sleep apnea or BP>140/90 will be excluded.
* Women with endometriosis and severe acute pain requiring immediate treatment will be excluded.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — women
Enrollment: 40 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Flow Mediated Vasodilation Microvascular skin blood flow analysis | 2 minutes
  Blood flow velocity will be measured using the Sonoscope S2 ultrasound imaging system.
Microdialysis perfusions | 15 minutes
  Following recovery from the microdialysis probe insertions we will measure resting skin blood flow (SkBF).

CONTACTS AND LOCATIONS:
Overall Officials: Nina Stachenfeld, MD, Principal Investigator — Yale University
Locations (1):
- Yale School of Medicine, New Haven, Connecticut, United States